CLINICAL TRIAL: NCT07223138
Title: A Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of Subcutaneous Sonelokimab in Participants With Psoriatic Arthritis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M1095-PSA-303; IZAR-OLE (Other: Sponsor)
Record Dates: First submitted 2025-10-20; First posted 2025-10-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
Keywords: Anti-Inflammatory Agents; Sonelokimab; Nanobody; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — sonelokimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: sonelokimab dose (Experimental): All participants will receive sonelokimab subcutaneously every 4 weeks
  Interventions: Drug: Sonelokimab

INTERVENTIONS:
Drug: Sonelokimab — Open-label

SUMMARY:
This is a study to demonstrate the long-term safety, tolerability and clinical efficacy of sonelokimab in the treatment of patients with psoriatic arthritis who completed a parental study (M1095-PSA-301 or M1095-PSA-302)

DETAILED DESCRIPTION:
M1095-PSA-303 is a Phase 3, multicenter, open-label extension study to investigate the long-term safety, tolerability and clinical efficacy of sonelokimab 60 mg subcutaneously every 4 weeks in patients with psoriatic arthritis who completed a parental study (M1095-PSA-301 or M1095-PSA-302).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who, in the opinion of the investigator, are expected to benefit from participation in this OLE study.
2. Participants who have received the second to last and/or last dose, as planned in the parental study, and have completed the end-of-treatment visit of the parental study.
3. Participants must have received their last dose of study treatment in the parental study no more than 8 weeks (but ideally 4 weeks) before the first dose in this OLE study.
4. Female participants are eligible to participate if they are not pregnant or breastfeeding and must be of nonchildbearing potential or must agree to use highly effective methods of contraception during the study and for at least 8 weeks after the last dose of study treatment. Female participant of childbearing potential must refrain from donating oocytes during the study and for at least 8 weeks after the last dose of study treatment.
5. Male participants must be willing to use a condom when sexually active with a partner of childbearing potential during the study and for at least 8 weeks after the last dose of study treatment, unless surgically sterile. Male participants must also agree to refrain from donating sperm during the study and for at least 8 weeks after the last dose of study treatment.

Exclusion Criteria:

1. Participants who met any of the discontinuation criteria of the parental study at the time of enrollment in this OLE study.
2. Participants who have ongoing or planned use of one or more of the prohibited PsA or non-PsA treatments specified in this protocol.
3. Participants who plan to participate in another interventional study for a drug or device during this study.
4. Participants who were unblinded during the parental study.
5. Participant noncompliance to the parental study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2028-02-04 (Estimated); Study Completion 2028-02-04 (Estimated)

PRIMARY OUTCOMES:
Long-term safety and tolerability of sonelokimab: | 52 weeks
  Treatment-emergent adverse events (TEAEs)
Long-term safety and tolerability of sonelokimab: | 52 weeks
  Serious adverse events (SAEs)
Long-term safety and tolerability of sonelokimab: | 52 weeks
  TEAEs leading to study withdrawal
Long-term safety and tolerability of sonelokimab: | 52 weeks
  Adverse events of special interest (AESIs)
Long-term safety and tolerability of sonelokimab: | 52 weeks
  Clinically significant changes in vital signs and standard 12-lead electrocardiogram Measure description: Number of participants with clinically significant changes in vital signs and 12-lead ECG intervals from baseline
Long-term safety and tolerability of sonelokimab: | 52 weeks
  Clinically significant changes in clinical laboratory parameters Measure description: Number of participants with clinically significant changes in hematology, biochemistry and urinalysis from baseline

SECONDARY OUTCOMES:
Long-term efficacy of sonelokimab: | 52 weeks
  Proportion of participants achieving American College of Rheumatology (ACR) 20/50/70% improvement criteria over time
Long-term efficacy of sonelokimab: | 52 weeks
  Change over time in Minimal disease activity (MDA)
Long-term efficacy of sonelokimab: | 52 weeks
  Change over time in Health assessment questionnaire-disability index (HAQ-DI)
Long-term efficacy of sonelokimab: | 52 weeks
  Change over time in Tender joint count (TJC)68/ swollen joint count (SJC)66
Long-term efficacy of sonelokimab: | 52 weeks
  Proportion of participants achieving Psoriasis Area and Severity Index (PASI) 75/90/100 over time
Long-term efficacy of sonelokimab: | 52 weeks
  Change over time in Modified Nail Psoriasis Severity Index (mNAPSI)
Long-term efficacy of sonelokimab: | 52 weeks
  Proportion of participants achieving Very low disease activity (VLDA) over time
Long-term efficacy of sonelokimab: | 52 weeks
  Proportion of participants achieving SpondyloArthritis Research Consortium of Canada (SPARCC) over time
Long-term efficacy of sonelokimab: | 52 weeks
  Change over time in Leeds Enthesitis Index (LEI)
Long term efficacy of sonelokimab | 52 weeks
  Proportion of participants achieving both an ACR 50/ACR70 and PASI90/100 improvement over time

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Site, Upland, California
  - Clinical Site, Duncansville, Pennsylvania
  - Clinical Site, Memphis, Tennessee